CLINICAL TRIAL: NCT03082495
Title: A Phase II Randomized Controlled Trial of Aerobic Exercise in Rectal Cancer Patients During and After Neoadjuvant Chemoradiotherapy
Brief Title: Exercise During and After Neoadjuvant Rectal Cancer Treatment
Acronym: EXERT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Canadian Cancer Society (CCS) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: HREBA.CC-16-0986
Record Dates: First submitted 2017-02-09; First posted 2017-03-17 (Actual); Last update posted 2022-05-27 (Actual); Status verified 2022-03

CONDITIONS: Rectal Cancer
Keywords: Exercise; Cancer; Symptom management; Quality of life; presurgical; chemoradiotherapy; Physical Fitness
MeSH Terms: conditions — Rectal Neoplasms; Motor Activity; Neoplasms | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor will be blinded to group assignment for the clinical outcomes including treatment toxicity, treatment completion, treatment response, and surgical complications.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise (Experimental): Aerobic exercise
  Interventions: Behavioral: Exercise
- Usual Care (No Intervention): Standard medical care

INTERVENTIONS:
Behavioral: Exercise — Supervised high-intensity interval training (HIIT) during NACRT followed by unsupervised moderate-to-vigorous intensity continuous exercise training after the completion of NACRT and before surgery
  Arms: Exercise

SUMMARY:
This study is designed to investigate if aerobic exercise during and after neoadjuvant chemoradiotherapy (NACRT) can improve outcomes for rectal cancer patients.

DETAILED DESCRIPTION:
The EXERT trial is a single-center, prospective, two-armed, phase II randomized controlled trial designed to test the preliminary efficacy of exercise training in this clinical setting and to further evaluate its feasibility and safety. Participants will be 60 rectal cancer patients scheduled to receive long-course NACRT followed by total mesorectal excision. Participants will be randomly assigned to exercise training or usual care. Participants in the exercise training group will be asked to complete three supervised, high-intensity interval training sessions/week during NACRT and ≥ 150 min/week of unsupervised, moderate-to-vigorous-intensity, continuous exercise training after NACRT prior to surgery. Participants in the usual care group will be asked not to increase their exercise from baseline. Assessments will be completed pre NACRT, post NACRT, and pre surgery. The primary endpoint will be cardiorespiratory fitness (VO2 peak) at the post-NACRT time point assessed by a graded exercise test. Secondary endpoints will include functional fitness, quality of life, and symptom management. Exploratory clinical endpoints will include treatment toxicities, treatment completion, treatment response, and surgical complications.

ELIGIBILITY:
Inclusion Criteria:

* All patients scheduled to receive long-course (5-6 weeks) of NACRT followed by total mesorectal excision

Exclusion Criteria:

* Unable to consent
* Unable to perform aerobic exercise
* Intention to engage in a structured exercise program during NACRT and/or after NACRT and prior to surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2017-06-26 (Actual); Primary Completion 2019-10-17 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
Change in Cardiorespiratory fitness | pre-NACRT (baseline), post-NACRT (an average of 6 weeks)
  VO2 peak

SECONDARY OUTCOMES:
Cardiorespiratory fitness | pre-surgery (an average of 12 weeks)
  VO2 peak
Functional fitness | pre-NACRT (baseline), post-NACRT (an average of 6 weeks), pre-surgery (an average of 12 weeks)
  Senior's Fitness Test
Generic quality of life | pre-NACRT (baseline), post-NACRT (an average of 6 weeks), pre-surgery (an average of 12 weeks)
  European Organisation for Research and Treatment of Cancer core 30-item questionnaire
Disease specific quality of life | pre-NACRT (baseline), post-NACRT (an average of 6 weeks), pre-surgery (an average of 12 weeks)
  European Organisation for Research and Treatment of Cancer questionnaire module for colorectal cancer
Symptom burden | pre-NACRT (baseline), post-NACRT (an average of 6 weeks), pre-surgery (an average of 12 weeks)
  M.D. Anderson Symptom Inventory
Exercise motivation | pre-NACRT (baseline), post-NACRT (an average of 6 weeks), pre-surgery (an average of 12 weeks)
  Theory of planned behaviour
Eligibility rate | up to 20 months
  Number of eligible patients divided by the number of rectal cancer patients scheduled to receive long-course NACRT
Recruitment rate | up to 20 months
  Number of patients randomized divided by the number of eligible patients
Exercise adherence rate | post-NACRT (an average of 6 weeks), pre-surgery (an average of 12 weeks)
  Exercise adherence during NACRT will be assessed by the number of exercise sessions attended out of 18 as well as adherence to the intensity and duration of the HIT intervals. Exercise adherence to the unsupervised exercise after NACRT will be assessed by self-report using the Godin Leisure-Time Exercise.
Follow-up assessment rate | post-NACRT (an average of 6 weeks), pre-surgery (an average of 12 weeks)
  Number of patients in each group completing the objective outcomes (cardiorespiratory fitness and functional fitness) and patient-reported outcomes (quality of life, symptom burden) at each timepoint.
Safety: Adverse event rate | post-NACRT (an average of 6 weeks), pre-surgery (an average of 12 weeks)
  Number of serious adverse events that occur during exercise testing or the supervised exercise sessions

OTHER OUTCOMES:
Treatment toxicities | every week during NACRT (up to 6 weeks)
  CTCAE Version 3.0
Number of patients completing 100% of their planned radiation dose within 1 week of planned completion date | post-NACRT (an average of 6 weeks)
  Obtained from electronic medical records
Number of patients receiving ≥ 80% of their planned chemotherapy dose | post-NACRT (an average of 6 weeks)
  Obtained from electronic medical records
Pathologic complete response rate | post-surgery (an average of 12 weeks)
  Obtained from electronic medical records
Length of hospital stay | post-surgery (an average of 12 weeks)
  Obtained from electronic medical records
Surgical approach | post-surgery (an average of 12 weeks)
  Obtained from electronic medical records
Ostomy | post-surgery (an average of 12 weeks)
  Obtained from electronic medical records
Sphincter preservation | post-surgery (an average of 12 weeks)
  Obtained from electronic medical records
Blood loss | post-surgery (an average of 12 weeks)
  Obtained from electronic medical records
Number of positive lymph nodes | post-surgery (an average of 12 weeks)
  Obtained from electronic medical records

CONTACTS AND LOCATIONS:
Overall Officials: Kerry S Courneya, PhD, Principal Investigator — University of Alberta
Locations (1):
- Cross Cancer Institute, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Morielli AR, Usmani N, Boule NG, Severin D, Tankel K, Joseph K, Nijjar T, Fairchild A, Courneya KS. Feasibility, Safety, and Preliminary Efficacy of Exercise During and After Neoadjuvant Rectal Cancer Treatment: A Phase II Randomized Controlled Trial. Clin Colorectal Cancer. 2021 Sep;20(3):216-226. doi: 10.1016/j.clcc.2021.05.004. Epub 2021 May 26. PMID 34158253
- [Background] Morielli AR, Boule NG, Usmani N, Tankel K, Joseph K, Severin D, Fairchild A, Nijjar T, Courneya KS. Effects of exercise during and after neoadjuvant chemoradiation on symptom burden and quality of life in rectal cancer patients: a phase II randomized controlled trial. J Cancer Surviv. 2023 Aug;17(4):1171-1183. doi: 10.1007/s11764-021-01149-w. Epub 2021 Nov 29. PMID 34841461
- [Derived] Arthuso FZ, Morielli AR, Usmani N, Joseph K, Nijjar T, Tankel K, Fairchild A, Severin D, Boule NG, Courneya KS. Effects of Exercise on Motivational Outcomes in Rectal Cancer Patients During and After Neoadjuvant Chemoradiation: A Phase II Randomized Controlled Trial. Semin Oncol Nurs. 2023 Aug;39(4):151419. doi: 10.1016/j.soncn.2023.151419. Epub 2023 Apr 13. PMID 37061361
- [Derived] Morielli AR, Usmani N, Boule NG, Severin D, Tankel K, Nijjar T, Joseph K, Fairchild A, Courneya KS. Exercise during and after neoadjuvant rectal cancer treatment (the EXERT trial): study protocol for a randomized controlled trial. Trials. 2018 Jan 12;19(1):35. doi: 10.1186/s13063-017-2398-1. PMID 29329555